CLINICAL TRIAL: NCT01793324
Title: Objective Assessment of Metabolic Monitoring in Patients Treated With Seroquel® or Seroquel® XR/Quetiapine Fumarate: Use of IMS Disease Analyzer to Assess Physician Behaviour in the UK and Germany
Brief Title: EMR Data to Assess Monitoring of Patients Treated With Quetiapine
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1443C00128
Record Dates: First submitted 2013-02-14; First posted 2013-02-15 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Schizophrenia; Bipolar Disorder; Major Depressive Disorder
Keywords: Effectiveness of risk minimization; Metabolic monitoring; Seroquel® or Seroquel® XR/quetiapine fumarate
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Depressive Disorder, Major

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GER: All patients with a diagnosis of schizophrenia, bipolar disorder or major depressive disorder treated with Seroquel® or Seroquel® XR seen by general practitioners and psychiatrists in Germany based upon patient encounters recorded in IMS Disease Analyzer during the calendar period 13 February 2012 - 31 August 2012
- UK: All patients with a diagnosis of schizophrenia, bipolar disorder or major depressive disorder treated with Seroquel® or Seroquel® XR seen by general practitioners in the United Kingdom based upon patient encounters recorded in IMS Disease Analyzer during the calendar period from 11 January 2012 - 31 July 2012

SUMMARY:
A study to evaluate the effectiveness of an update of educational materials with respect to evaluation of monitoring of metabolic parameters

DETAILED DESCRIPTION:
Objective assessment of metabolic monitoring in patients treated with Seroquel® or Seroquel® XR/quetiapine fumarate: use of IMS Disease Analyzer to assess physician behaviour in the UK and Germany

ELIGIBILITY:
Inclusion Criteria:

- Electronic medical records of patients with diagnoses of schizophrenia, Bipolar Disorder (BPD) or Major Depressive Disorder (MDD) treated with Seroquel® or Seroquel®XR during the calendar periods: 13 Feb - 31 Aug 2012 seen by GP & psychiatrists in Germany & 11 Jan-31 July 2012 seen by GPs in the UK

Exclusion Criteria:

- Patients with above mentioned diagnoses treated with Seroquel® or Seroquel® XR/quetiapine fumarate not having any medical encounters during the time periods: 13 Feb - 31 Aug 2012 in Germany & 11 Jan-31 July 2012 by GPs in the UK

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cross sectional assessment of physician encounters with patients
Sampling Method: Non-Probability Sample
Enrollment: 6153 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Determination whether physicians in the UK and Germany perform monitoring of patients treated with Seroquel® and Seroquel® XR including measurement of the following during patient encounters: weight at drug initiation and over the course of treatment. | Over 6 months following the distribution of metabolic educational materials in the country
Monitoring of hyperlipidemia during patient encounters. | Over 6 months following the distribution of metabolic educational materials in the country
Monitoring for signs and symptoms of hyperglycemia during patient encounters. | Over 6 months following the distribution of metabolic educational materials in the country
Monitoring of blood glucose in patients with diabetes; monitoring of patients with risk factors for diabetes for worsening of glycemic control during patient encounters. | Over 6 months following the distribution of metabolic educational materials in the country
Counseling patients on healthy eating, exercise and healthy lifestyle improvements during patient encounters. | Over 6 months following the distribution of metabolic educational materials in the country

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Brody, MPH, Principal Investigator — AZ